CLINICAL TRIAL: NCT04992338
Title: Pilot Study to Analyze the Effects of the Use of the Mobile Application CarpeDiem (Collaborative and Adaptive Recommender for PersonalizedDIEtManagement) on Lifestyle Habits
Brief Title: Collaborative and Adaptive Recommender for Personalized DIEt Management
Acronym: CarpeDiem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2
Record Dates: First submitted 2021-07-21; First posted 2021-08-05 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Diet Habit; Sleep; Life Style, Healthy; Physical Activity
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - CarpeDiem app (Experimental): Participants will receive at their home the activity tracker of Fitbit brand, model Inspire HR 2, as well as instructions to download and use the CarpeDiem application and the Fitbit application in their mobile phones and synchronize the bracelet. The intervention consists of detecting unhealthy user behaviors and, through contextualized and personalized recommendations and strategies based on gamification, modifying said behaviors and motivating individuals to maintain this modification over time in order to prevent illnesses associated with bad habits. The intervention is performed through the CarpeDiem application, participants will be able to answer follow-up questionnaires, carry out missions designed to improve their eating habits, monitor their physical activity and sleep.
  Interventions: Device: Mobile app
- Control group - Activity tracker + general recommendations (No Intervention): Participants will receive the Fitbit activity tracker, model Inspire HR 2. They will also receive instructions to download the Fitbit application from their mobile phone and synchronize the bracelet. Additionally, this group will receive general recommendations on healthy lifestyle habits through standardized documents that contain general guidelines, such as: "Get in the habit of going to sleep and always waking up at the same time, even on weekends."

INTERVENTIONS:
Device: Mobile app — The CarpeDiem application is a mobile application, designed in collaboration with the Health and Nutrition Technology Unit (UTNS, Eurecat) and the translational research group on respiratory medicine of the Institut de Recerca Biomèdica de Lleida. The application is available for devices with Android as the operative system and its advanced interface allows the user to monitor their physical activity, sleep and diet and motivate them to meet personalized goals through gamification. To do this, the user must answer the questionnaires that they will find on the main page of the application with a predetermined frequency, as well as perform missions that will help them acquire healthier habits. In addition, the user will receive motivational messages and recommendations through notifications that will help and guide them to achieve their missions and achieve their goals, and as a result of changing habits.
  Arms: Intervention group - CarpeDiem app

SUMMARY:
CarpeDiem is a mobile application which provides personalized and holistic recommendations in the area of diet, physical activity and sleep to help their users adopt a healthier lifestyle. In this study it is hypothesized that the usage of this application can achieve a more effective lifestyle improvement than an intervention with the use of wearables, their respective generic applications and general healthy lifestyle recommendations. Therefore, this study aims to assess whether the incorporation of a mobile application such as CarpeDiem, which includes smart, personalized and holistic recommendations related to a healthy lifestyle (diet, physical activity and sleep) is associated with a more pronounced change in healthy lifestyle habits than a passive monitoring approach using wearables and the administration of general recommendations.

This clinical trial consists of a multicenter pilot study performed at the headquarters of the Technology Center of Catalonia (Eurecat), randomized, parallel and controlled, performed with healthy adults (18 to 65 years old). 100 subjects will be recruited, 50 as an intervention group and 50 as a control group. The study is scheduled to begin in June 2021.

Both groups will receive an activity tracker (Fitbit Inspire HR 2). The intervention group will also receive instructions to download and use the CarpeDiem application. Through the CarpeDiem application, participants will be able to answer follow-up questionnaires, perform missions related to the healthy consumption of various food groups, monitor their physical activity and sleep, and receive periodic, personalized and holistic recommendations based on the three pillars of health. The control group will receive instructions to download the Fitbit application and will additionally receive general recommendations for healthy lifestyle habits through standardized documents. Both groups will be provided access to the initial and final questionnaires that will be done online. All participants must return the signed informed consent either with a digital signature or by mail to the Eurecat-Barcelona headquarters.

The main variable of the study is: the Mediterranean lifestyle index, calculated from the short MEDLIFE questionnaire with 28 items, validated for the Spanish adult population.

The secondary variables are:

Diet related: Food intake and food groups taken from the Food Frequency Questionnaire (CFCA). Diet diversity index calculated from the CFCA.

Related to physical activity: Total physical activity in MET-minutes / week, extracted from the IPAQ questionnaire. Data referring to daily activity (minutes sitting and moderate and intense physical activity and number of steps taken) measured with the activity bracelet.

Sleep-related: Sleep quality index, derived from the Pittsburg Sleep Quality Questionnaire (PSQI). Data referring to users' daily sleep (sleep duration, efficiency, start and end) measured with the activity bracelet.

Related to the user's experience in using the application, evaluated through the UEQ questionnaire. Only at the end of the intervention.

In total, subjects will receive 3 visits:

Visit 0, pre-screening visit before randomization to check inclusion / exclusion criteria, using an online form.

Visit 1, after randomization, inclusion visit. Participants will receive the activity bracelet and informed consent at their homes. During this visit, participants will answer the questionnaires using online forms.

Visit 2, after three months, final visit of the study intervention. Participants will answer the questionnaires using online forms.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are between 18 and 65 years old.
* Owners of a smartphone or tablet with Android 6.0 operative system version or higher (API 23), with internet access and Bluetooth connectivity.
* Must accept the informed consent .

Exclusion Criteria:

* Pregnancy or lactation
* Having a physical limitation to perform physical activity
* Usage of another app to monitor their lifestyle habits (nutrition, physical activity or sleep)
* Have a diagnosed sleep disorder or are taking sleep medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-11-28 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Mediterranean Lifestyle Index, (MEDLIFE) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Eurecat, Reus, Spain

IPD SHARING:
Plan to Share IPD: No